CLINICAL TRIAL: NCT07354581
Title: Comparison of Ultrasound-Guided Erector Spinae Plane Block and Quadro-Iliac Plane Block for Postoperative Analgesia Management Following Lumbar Instrumentation Surgery
Brief Title: Erector Spinae Plane Block vs Quadro-Iliac Plane Block After Lumbar Instrumentation Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Merih Yıldız Eglen, principal investigator,MD, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BursaCity Hos 2
Record Dates: First submitted 2025-12-31; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative
Keywords: Lumbar instrumentation; Postoperative pain management; Erector Spinae Block; Quadro-Iliac Plane Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (ESPB) (Active Comparator): Participants in this arm will receive an ultrasound-guided Erector Spinae Plane Block at the end of surgery, before extubation, with the patient in the prone position under standard sterilization conditions. The block will be performed bilaterally as part of a standardized multimodal postoperative analgesia protocol following lumbar instrumentation surgery.
  Interventions: Procedure: Erector Spinae Plane Block
- Quadro-Iliac Plane Block (QIPB) (Active Comparator): Participants in this arm will receive an ultrasound-guided Quadro-Iliac Plane Block at the end of surgery, before extubation, with the patient in the prone position under standard sterilization conditions. The block will be performed bilaterally as part of a standardized multimodal postoperative analgesia protocol following lumbar instrumentation surgery.
  Interventions: Procedure: Quadro-Iliac Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — An ultrasound-guided Erector Spinae Plane Block will be performed at the end of surgery, before extubation, with the patient in the prone position under standard sterilization conditions. The ultrasound probe will be placed in the parasagittal plane at the level corresponding to the surgical site to visualize the transverse process and erector spinae muscle. Following confirmation of correct needle placement with 2 mL of normal saline, 20 mL of 0.25% bupivacaine will be injected into the fascial plane deep to the erector spinae muscle. The block will be performed bilaterally, with a total volume of 40 mL, as part of a standardized multimodal postoperative analgesia protocol.
  Arms: Erector Spinae Plane Block (ESPB)
Procedure: Quadro-Iliac Plane Block — An ultrasound-guided Quadro-Iliac Plane Block will be performed at the end of surgery, before extubation, with the patient in the prone position under standard sterilization conditions. A convex ultrasound probe will be placed at the level where the quadratus lumborum muscle attaches to the iliac crest to visualize the erector spinae muscle and the underlying quadratus lumborum muscle. The block location will be confirmed with the injection of 2 mL of isotonic solution, followed by the injection of 20 mL of 0.25% bupivacaine. The spread of the local anesthetic between the erector spinae muscle and quadratus lumborum muscle will be observed under ultrasound guidance. The block will be performed bilaterally, with a total volume of 40 mL, as part of a standardized multimodal postoperative analgesia protocol.
  Arms: Quadro-Iliac Plane Block (QIPB)

SUMMARY:
Lumbar instrumentation surgery is associated with significant postoperative pain. This study compares the postoperative analgesic effectiveness of ultrasound-guided Erector Spinae Plane Block and Quadro-Iliac Plane Block in patients undergoing lumbar instrumentation surgery.

DETAILED DESCRIPTION:
Lumbar instrumentation surgery is frequently associated with moderate to severe postoperative pain, which may negatively affect patient comfort, delay mobilization, and increase opioid consumption. Effective postoperative analgesia is therefore essential for improving recovery and reducing opioid-related adverse effects. Regional anesthesia techniques have become an important component of multimodal analgesia strategies in lumbar spine surgery.

The Erector Spinae Plane Block (ESPB) is a well-established ultrasound-guided regional anesthesia technique that has been shown to provide postoperative analgesia in various spinal procedures. The Quadro-Iliac Plane Block (QIPB) is a newly developed ultrasound-guided block targeting the fascial plane between the erector spinae muscle and the quadratus lumborum muscle at the level of the iliac crest, with the potential to provide effective analgesia for lumbar spine surgeries. However, comparative clinical data regarding the analgesic effectiveness of these two techniques in lumbar instrumentation surgery are limited.

This study is designed to compare the postoperative analgesic effectiveness of ultrasound-guided ESPB and QIPB in patients undergoing elective lumbar instrumentation surgery under general anesthesia. Both blocks will be performed using ultrasound guidance as part of a standardized multimodal analgesia protocol.

The findings of this study aim to clarify the relative effectiveness of ESPB and QIPB for postoperative pain control following lumbar instrumentation surgery and to contribute to evidence-based selection of regional analgesia techniques in lumbar spine procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Classified as American Society of Anesthesiologists physical status I-III
* Scheduled for elective lumbar instrumentation surgery under general anesthesia
* Provision of written informed consent

Exclusion Criteria:

* Use of anticoagulant medications or presence of bleeding diathesis
* Known allergy or hypersensitivity to local anesthetics or opioid drugs
* Infection at the planned block site
* Alcohol or drug dependence
* Cognitive impairment preventing reliable pain assessment
* Pregnancy or lactation
* History of previous lumbar spine surgery
* Diabetes mellitus
* Renal or hepatic insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative 48-Hour PCA Opioid Consumption | Postoperative 0-8, 8-16, 16-24, 24-48 intervals
  Total amount of opioid delivered by the patient-controlled analgesia (PCA) device during the first 48 hours after surgery, recorded in milligrams (mg).

SECONDARY OUTCOMES:
QoR-15 Recovery Score | Postoperative 24th and 48th hours
  The investigators will use the Turkish version of Quality of Recovery (QoR) / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  Able to breathe easily Been able to enjoy food Feeling rested Have had a good sleep Able to look after personal toilet and hygiene unaided Able to communicate with Getting support from hospital doctors and nurses Able to return to work or usual home activities Feeling comfortable and in control Having a feeling of general well-being
  PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) Moderate pain Severe pain Nausea or vomiting Feeling worried or anxious Feeling sad or depressed
Dynamic and static Numeric Rating Scale scores | 0, 2, 4, 8, 16, 24, and 48 hours postoperatively]
  Numeric Rating Scale (NRS) (0-10; 0= no pain, 10= the most severe pain felt ) pain scores at rest or movement at predefined postoperative hours
Total rescue analgesic dose | Postoperative 24th and 48th hours
  Despite the use of patient-controlled analgesia (PCA), if the Numeric Rating Scale (NRS) score is ≥4 at any time point, 0.5 mg/kg intravenous meperidine will be administered as rescue analgesia.
  Total amount of meperidin during the first 24 and 48 hours after surgery, recorded in milligrams (mg).
Time of first request for rescue analgesia | Postoperative 48 hours
  Despite the use of patient-controlled analgesia (PCA), if the Numeric Rating Scale (NRS) score is ≥4 at any time point, 0.5 mg/kg intravenous meperidine will be administered as rescue analgesia.
Length of Hospital Stay | The time from the end of the surgery to discharge from the hospital(day)
  Length of hospital stay will be defined as the number of days from the end of surgery to hospital discharge.
Block and Opioid-Related Adverse Effects and Complications | Postoperative 48 hours
  Block- and opioid-related adverse effects and complications, including but not limited to local anesthetic toxicity, hematoma, infection, nerve injury, nausea, vomiting, pruritus, sedation, and respiratory depression, will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Girit M, Akin T, Narayanan M, Alici HA. Ultrasound guided quadro-iliac plane block: another novel fascial plane block. Pain Med. 2024 May 3;25(6):370-373. doi: 10.1093/pm/pnae018. PMID 38459608
- [Result] Turan EI, Sahin AS. Quadro-iliac plane block (QIPB) in lumbar stabilisation surgeries: A case series. Indian J Anaesth. 2025 Feb;69(2):244-245. doi: 10.4103/ija.ija_1077_24. Epub 2025 Jan 29. No abstract available. PMID 40160919
- [Result] Ciftci B, Cetinkal A, Alver S, Ahiskalioglu A. Quadro-iliac plane block for lumbar multi-level instrumentation surgery: far away from the surgical area. Minerva Anestesiol. 2025 Apr;91(4):358-359. doi: 10.23736/S0375-9393.24.18680-4. Epub 2024 Dec 10. No abstract available. PMID 39656149